CLINICAL TRIAL: NCT05616468
Title: Clinical Study of the Safety and Initial Efficacy of BGT007 Cells in the Treatment of Patients With Relapsed /Metastatic Nasopharyngeal Carcinoma
Brief Title: BGT007 Cell Treatment of Nasopharyngeal Carcinoma
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Hospital of Xuzhou Medical University (Other)
Collaborators: Guangzhou Bioresette Biomedical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BR-BGT-001
Record Dates: First submitted 2022-10-30; First posted 2022-11-15 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: CAR-T; nasopharyngeal carcinoma; recurrent/metastatic nasopharyngeal carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — fludarabine; fludarabine phosphate; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BGT007 Cell Injection (Experimental): In this study, 23 patients diagnosed with recurrent/metastatic nasopharyngeal carcinoma will receive a single intravenous infusion of BGT007 cells after enrollment, with a dose of 5.0 × 10^5cells/kg，1.0 × 10^6cells/kg，3.0 × 10^6cells/kg，6.0 × 10^6cells/kg，1.0 × 10^7cells/kg。 One subject was enrolled in each of the first two dose groups, and the other three dose groups were enrolled in accordance with the conventional "3+3" dose increase.
  Interventions: Biological: BGT007 Cell Injection; Drug: Fludarabine; Drug: cyclophosphamide

INTERVENTIONS:
Biological: BGT007 Cell Injection — BGT007 cells (d0) were infused intravenously once, and the dose group was 5.0 × 10^5cells/kg，1.0 × 10^6cells/kg，3.0 × 10^6cells/kg，6.0 × 10^6cells/kg，1.0 × 10^7cells/kg。
Drug: Fludarabine — Fludarabine 25~30mg/m2/d was infused intravenously for 3 consecutive days. (- 5 days to - 3 days)
  Other Names: FLUDARA
Drug: cyclophosphamide — 250~350mg/m2/d cyclophosphamide was infused intravenously for 3 consecutive days. (- 5 days to - 3 days)
  Other Names: Cytoxan

SUMMARY:
This is an exploratory study to evaluate the safety and preliminary effectiveness of BGT007 cells in the treatment of recurrent/metastatic nasopharyngeal carcinoma

DETAILED DESCRIPTION:
The researchers designed a single arm, open, exploratory study to improve the "3+3" dose escalation. The maximum dose or the best effective dose shall be determined according to the subject and dose increasing test to verify the safe and effective number of cells per unit weight. The improved "3+3" dose increasing design was adopted, and BGT007 cells were set with 5 dose groups that were gradually increased for treatment evaluation. The dose groups were 5.0 × 10^5cells/kg，1.0 × 10^6cells/kg，3.0 × 10^6cells/kg，6.0 × 10^6cells/kg，1.0 × 10^7cells/kg。 Cell reinfusion will be carried out on day 0 (d0), and each subject will be observed for at least 4 weeks after receiving cell reinfusion (DLT observation period)

ELIGIBILITY:
Inclusion Criteria:

* 1. Sign the written informed consent voluntarily;
* 2. Age ≥ 18, ≤ 75, male or female;
* 3.Expected life ≥ 3 months
* 4. The physical condition score of the Eastern Tumor Cooperative Organization (ECOG) is 0-2;
* 5.Biopsy sample or pathological wax slice test (within 1 year before signing the informed consent): target test positive
* 6. According to RECIST v1.1 solid tumor evaluation criteria, there is at least one measurable lesion;
* 7. Patients with recurrent/metastatic nasopharyngeal carcinoma who have received second-line or above system treatment failure in the past (Recurrence of nasopharyngeal carcinoma: nasopharyngeal carcinoma confirmed by pathology, after radical radiotherapy, the clinical tumor disappears completely, and after 6 months of treatment, local tumors with the same pathological type as the original tumor reappear; metastasis of nasopharyngeal carcinoma: tumor cells transfer from the primary site to distant organs through various ways, such as blood and lymph, and form tumor metastasis focus);
* 8. It is possible to establish a single blood collection or venous blood collection channel, and there is no other blood cell separation contraindication;
* 9. It has sufficient organ and bone marrow functions, as defined below

routine blood test

Neutrophil count (NEUT #) ≥ 1.0 × 10^9/L

Platelet count (PLT) ≥ 80 × 10^9/L

Hemoglobin concentration ≥ 90g/L

Liver function: subjects without liver metastasis

Aspartate aminotransferase (AST) ≤ 2.5 × Upper limit of normal value (ULN)

Alanine aminotransferase (ALT) ≤ 2.5 × Upper limit of normal value (ULN)

Total bilirubin (TBIL) ≤ 1.5 × ULN

Liver function: subjects with liver metastasis

Aspartate aminotransferase (AST) ≤ 5 × Upper limit of normal value (ULN)

Alanine aminotransferase (ALT) ≤ 5 × Upper limit of normal value (ULN)

Liver function: subjects with liver metastasis or Gilbert syndrome

Total bilirubin (TBIL) ≤ 2 × ULN

renal function

Creatinine clearance rate (CCR) ≥ 50mL/min

Coagulation function

International normalized ratio (INR) ≤ 1.5 × ULN

Activated partial thromboplastin event (APTT) ≤ 1.5 × ULN

* 10. Toxic side effects left by early anti-tumor therapy (radiotherapy, chemotherapy, targeted therapy, etc.) ≤ Level 1 (CTCAE5.0);
* 11. During the study period and within 6 months after the last administration, subjects with fertility (male or female) must take effective medical contraceptive measures. Female subjects of childbearing age must have a pregnancy test within 72 hours before the first administration, and the result is negative.

Exclusion Criteria:

* 1. Active central nervous system metastasis (except those that are stable after treatment);
* 2. HIV positive or HBsAg positive, HBV DNA copy number is positive (quantitative test ≥ 1000 cps/ml) or HCV antibody is positive and HCV RNA is positive;
* 3. Those who have mental or psychological diseases and cannot cooperate with the treatment and efficacy evaluation;
* 4. Subjects with severe autoimmune diseases and long-term application of immunosuppressants;
* 5. There is active infection or uncontrollable infection requiring systemic treatment within 14 days before signing the informed consent form;
* 6. Any unstable systemic disease (including but not limited to): Active infection (except local infection);

Unstable angina pectoris;

Cerebrovascular ischemia or cerebrovascular accident (within 6 months before screening);

Myocardial infarction (within 6 months before screening);

Congestive heart failure (New York Heart Association [HYHA] classification ≥ Ⅲ);

Serious arrhythmia requiring drug treatment;

Heart disease needs treatment or hypertension is out of control after treatment (blood pressure>160mmHg/100mmHg);

* 7. Complicated with dysfunction of lung, brain, kidney and other important organs;
* 8. Subjects had undergone major surgery or severe trauma within 4 weeks before signing the informed consent form, or were expected to undergo major surgery during the study period.
* 9. Subjects received the last radiotherapy or anti-tumor treatment (chemotherapy, targeted therapy or immunotherapy) within 4 weeks before signing the informed consent form;
* 10. The subject currently suffers from or has suffered from other malignant tumors that cannot be cured within 3 years, except for cervical cancer or skin basal cell cancer, and other malignant tumors with a disease-free survival period of more than 5 years;
* 11. Have received T cells (including CAR-T and TCR-T) modified by chimeric antigen receptor within half a year before signing the informed consent form;
* 12. Graft versus host disease (GVHD)
* 13. Subjects who were receiving systemic steroid treatment before signing the informed consent form and who were judged by the investigator to need long-term use of systemic steroid treatment during the treatment period (except for inhalation or local use); And subjects treated with systemic steroids within 72 hours before cell reinfusion (except for inhalation or local use);
* 14. Serious allergy or allergy history
* 15. Subjects requiring anticoagulation treatment
* 16. Pregnant or lactating women, or have a pregnancy plan within six months (for both men and women);
* 17. The investigator believes that there are other reasons that cannot be included in the treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2022-12-30 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity（DLT） | From day 0 to day 28
  Adverse events related to cell therapy were observed on 28 days after BGT007 cell injection , as specified in the protocol

SECONDARY OUTCOMES:
Cmax | 12 months
  The amplification of BGT007 cells in peripheral blood peaked after administration
Tmax | 12 months
  Number of days of peak BGT007 cell expansion after administration
AUC(Day 0 to Day 28) | From day 0 to day 28
  The area under the curve of BGT007 cells from day 0 to day 28 after administration was plotted by the visit time of BGT007 cells in peripheral blood
ORR | 12 months
  Proportion of patients who achieved pre-defined tumor volume reduction and maintained the minimum time limit.Imaging examination was performed after administration, and RECIST1.1 evaluation criteria was used for evaluation
PFS | 12 months
  The time from the onset of leukocyte apheresis to the appearance of tumor progression or death.
OS | 12 months
  The time between leukocyte apheresis and death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu, China